CLINICAL TRIAL: NCT06948734
Title: Longitudinal Monitoring of Pulpal and Periapical Health of Adjacent Natural Teeth Before and After Implant Placement
Brief Title: Longitudinal Assessment of Adjacent Tooth Health Following Implant Placement
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Helin Kussever, Research Assistant, Cukurova University
Other Study IDs: 2023/134/53
Record Dates: First submitted 2025-04-18; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-11

CONDITIONS: Dental Implants; Postoperative Period; Endodontics; Health
Keywords: Dental implants; Postoperative monitoring; Adjacent teeth; Pulpal health
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for implant placement in edentulous sites adjacent to natural teeth: Patients scheduled to receive multiple implants at different time points, in edentulous sites adjacent to natural teeth, based on individualized surgical planning.
  Interventions: Diagnostic Test: Clinical and radiographic examination

INTERVENTIONS:
Diagnostic Test: Clinical and radiographic examination — In order to evaluate the pulpal and periapical health of natural teeth adjacent to dental implants at specific time intervals, percussion, palpation, and pulpal diagnostic tests were performed, and the presence of any pathological changes was monitored using radiographic examinations.

SUMMARY:
This study is a cohort investigation involving patients scheduled to receive dental implants in edentulous sites adjacent to natural teeth. Individuals aged between 18 and 65 years, without any systemic diseases and possessing natural teeth adjacent to the planned implant sites, were included. Clinical and radiographic evaluations were conducted preoperatively, and at 1 week, 1 month, and 3 months following implant placement. The null hypotheses (H0) of this study are as follows: First, there is no significant difference in the clinical parameters of adjacent teeth before and after implant surgery. Second, there is no significant change in the radiological parameters in adjacent teeth between the preoperative and postoperative periods.

DETAILED DESCRIPTION:
Modern implantology began in 1965 with the placement of four intraosseous titanium implants in a patient with a mandibular defect, marking the introduction of the concept of osseointegration. Since then, dental implants have emerged as a reliable and effective treatment modality for the rehabilitation of edentulous spaces. This longitudinal cohort study aims to evaluate whether dental implants placed in edentulous sites adjacent to natural teeth lead to alterations in the endodontic condition of these neighboring teeth. Specifically, the study investigates the nature and extent of any pulpal or periapical changes in adjacent teeth following implant placement. It is hypothesized that any damage to the adjacent teeth may be attributed to intraoperative complications, iatrogenic factors, or physiological consequences associated with the healing of hard and soft tissues post-surgery. The short-term observation intervals (1 week, 1 month, and 3 months postoperatively) are expected to offer insights into the potential causes of endodontic symptoms that may arise in neighboring teeth. Through this design, the study seeks to better understand the etiological relationship between implant placement and the pulpal/periapical health of adjacent teeth.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years ASA I or II classification At least one vital adjacent tooth at implant site Adjacent tooth free of pulpal/periapical pathology Not prosthetically restored; unrestored or restored with composite material Sites allowing a tooth-implant distance of ≥1.5 mm Patients scheduled to receive multiple implants at different time points based on surgical planning

Exclusion Criteria:

Age <18 or >65 ASA physical status classification ≥ III Absence of adjacent teeth at implant site Undergoing or planned advanced implant procedures (e.g., bone grafting, sinus lifting, nerve lateralization/transposition) Adjacent teeth devital, with periapical pathology, root canal treated, or prosthetically rehabilitated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 65 years, without any systemic diseases, who were scheduled to receive multiple dental implants at different time points in edentulous sites adjacent to natural teeth, based on individualized surgical planning
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Percussion and Pulpal Diagnostic Test Outcomes | At the preoperative stage and during postoperative follow-ups at 1 week, 1 month, and 3 months the tests were performed.
  At the preoperative stage and during postoperative follow-ups at 1 week, 1 month, and 3 months, vertical percussion was performed on the natural teeth adjacent to the dental implant by gently placing a dental probe under its own weight. The response was recorded as either positive or negative. Electric pulp test and cold test (pulpal diagnostic tests) were also performed on the adjacent teeth at the same time intervals. Numerical responses were recorded for the electric pulp test, while responses to the cold test were documented as either positive or negative.
Palpation Test Outcomes | At the preoperative stage and during postoperative follow-ups at 1 week, 1 month, and 3 months the tests were performed.
  To assess the presence or absence of tenderness upon palpation, a bidigital palpation test was performed during the preoperative phase and at postoperative follow-up visits at 1 week, 1 month, and 3 months. The response was recorded as either positive or negative.
Measurement of pain scores using the Numeric Pain Rating Scale (NPRS) | At the preoperative stage and during postoperative follow-ups at 1 week, 1 month, and 3 months the tests were performed.
  At the preoperative stage and during postoperative follow-ups at 1 week, 1 month, and 3 months, patients were asked to indicate the number corresponding to the intensity of pain they experienced on a 0-10 Numerical Rating Scale (NRS), and the selected values were recorded.
Assessment of Radiological Outcomes | At the preoperative stage and during postoperative follow-up at 3 months the tests were performed.
  Periapical status of the natural teeth adjacent to the dental implants was assessed radiographically at baseline and at the 3-month postoperative follow-up. Radiographs were evaluated for the presence of any periapical pathology, and outcomes were documented as either 'radiolucent area present' or 'radiolucent area absent'.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University Faculty of Dentistry Department of Endodontics, Adana, Sarıcam, Turkey (Türkiye)